CLINICAL TRIAL: NCT00225342
Title: Effects of Rosiglitazone and Sulphonylureas on Ischaemic Burden, Blood Pressure and Novel Risk Markers Inclusive of Vascular Function in Patients With Chronic Stable Angina and Type 2 Diabetes Mellitus: A Randomised, Double-Blinded Study.
Brief Title: Study Protocol for Rosiglitazone Versus Gliclazide in Diabetics With Angina
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GlasUniRosiGlic; Eudract No. 2004-000943-40
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Angina Pectoris; Diabetes Mellitus, Type 2
Keywords: Angina; Ischaemic heart disease; Diabetes
MeSH Terms: conditions — Angina Pectoris; Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus | interventions — Rosiglitazone; Gliclazide

INTERVENTIONS:
Drug: Rosiglitazone
Drug: Gliclazide (Comparison drug)

SUMMARY:
The principle objective of the trial is to compare rosiglitazone to gliclazide in patients with type 2 diabetes mellitus and chronic stable angina to see how the subjects' angina status changes.

Angina status will be measured via exercise tolerance testing, 24-hour ECG testing and angina quality of life questionnaire.

DETAILED DESCRIPTION:
Ischaemic heart disease is one of the main complications of type 2 diabetes mellitus, both in terms of morbidity and mortality. Reducing plasma glucose with hypoglycaemic agents has not been shown to improve cardiovascular mortality or morbidity. Chronic stable angina is a common problem in patients with type 2 diabetes mellitus.

We postulate that in subjects with uncontrolled type 2 diabetes mellitus (Hba1c >7.5%), on metformin therapy, and chronic stable angina that the addition of the insulin sensitiser, rosiglitazone to control their diabetes will improve their angina when compared to the addition of the hypoglycaemic agent gliclazide. This hypothesis is based on the fact that insulin resistance is an upstream mechanism common to both conditions.

We will randomise such patients to 3 months therapy of rosiglitazone or gliclazide for 3 months, comparing angina status before and after by way of full Bruce protocol exercise testing, 24 hour ST segment analysis and angina questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable angina with ongoing symptoms. (The treatment goal being an improvement in symptoms)
* Participants will have uncontrolled diabetes (Hba1c>7.5) on metformin monotherapy (so the diabetes is not over treated)
* Participants will be diabetic for less than 8 years.

Exclusion Criteria:

* Renal impairment (creatinine >130mmol/l)
* Hepatic Impairment (ALT>70U/l, AST>80U/l)
* Any clinical signs of heart failure
* Physical disability precluding treadmill exercise tolerance testing
* Abnormal resting ECG (left or right bundle-branch block, left or right ventricular hypertrophy, ventricular preexcitation, Q-wave myocardial infarction, digitalis therapy)
* Women of childbearing potential
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
Angina status at 3 months

SECONDARY OUTCOMES:
Pulse wave velocity at 3 months
Small vessel function at 3 months
Haemostatic markers at 3 months
Biochemical markers of inflammation at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Sattar, MBChB PhD, Principal Investigator — University of Glasgow; Stuart M Cobbe, MBChB MD, Principal Investigator — University of Glasgow
Locations (1):
- Cardiology Department, Glasgow Royal Infirmary, Glasgow, United Kingdom